CLINICAL TRIAL: NCT06888063
Title: Preventing Liver Recurrence After Partial Hepatectomy for Intrahepatic Cholangiocarcinoma Using Adjuvant Hepatic Arterial Infusion Pump Chemotherapy - PUMP IV Trial
Brief Title: Additional Chemotherapy Administered Directly Into the Liver Using a Chemo Pump in Patients With Bile Duct Cancer Inside the Liver Treatable by Surgery
Acronym: PUMP IV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Koningin Wilhelmina Fonds (Other)
Responsible Party: Principal Investigator, Bas Groot Koerkamp, MD, PhD, Principal Investigator and Professor of Pancreato-Biliary Surgery, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2024-0324; 2024-513726-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-05; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Intrahepatic Bile Duct Cancer; Intrahepatic Cholangiocarcinoma (Icc); Intrahepatic Bile Duct Carcinoma; Intrahepatic Cholangiocarcinoma
Keywords: PUMP; PUMP IV; Hepatic Arterial Infusion Chemotherapy; Hepatic Arterial Infusion Pump chemotherapy; HAIP; HAIC; Intrahepatic cholangiocarcinoma; iCCA; Floxuridin; Chemopump
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension | interventions — Floxuridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Surgery + chemo pump (Hepatic Arterial Infusion Pump chemotherapy) (Experimental): Surgery + chemo pump
  Interventions: Combination Product: Hepatic Arterial Infusion Pump chemotherapy with floxuridin

INTERVENTIONS:
Combination Product: Hepatic Arterial Infusion Pump chemotherapy with floxuridin — Participants in this arm will receive in addition to standard care (surgery) a chemo pump. This pump will provide participants with 4 cycles of treatment with chemotherapy (Floxuridin), each lasting 4 weeks. Total treatment with chemotherapy will last 16 weeks (approx. 4 months)
  Other Names: HAIP; HAIC with floxuridin; PUMP chemotherapy

SUMMARY:
The goal of this clinical trial is to learn if additional chemotherapy by means of a chemo pump can prevent return of disease in adult patients with bile duct cancer in the liver that can be treated with surgery. The main questions it aims to answer are:

* Does addition of chemotherapy by means of a chemo pump lead to less return of disease within the liver two years after surgery?
* Does addition of chemotherapy by means of a chemo pump lead to longer survival of patients?
* Does addition of chemotherapy by means of a chemo pump lead to an increase in quality of life?

Participants will receive an implanted chemo pump, through which additional chemotherapy will be given to the liver in addition to surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* ECOG or WHO performance status 0 or 1
* Diagnosis of resectable iCCA on imaging. No histological confirmation is needed before surgery, according to standard of care.
* Patient is able to undergo a laparotomy.
* Positioning of a catheter for HAIP chemotherapy is technically feasible based on a CT-scan with early arterial phase with 1mm cuts. The default site for the catheter insertion is the GDA. Accessory or aberrant hepatic arteries are no contraindication for catheter placement.
* Adequate bone marrow, liver, and renal function before inclusion (values may be max. 30 days old)
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^ 9/L
* White blood cell count (WBC) ≥ 2.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Glomerular filtration rate (GFR) ≥ 30 ml/min
* Haemoglobin (Hb) ≥ 5.5 mmol/L
* Total bilirubin ≤ 25 µmol/L
* Written informed consent must be given according to ICH/good clinical practice (GCP), and national/local regulations.

Exclusion Criteria:

* Presence of extrahepatic disease at the time of first presentation. Patients with locoregional lymph node disease or with small (≤ 1 cm) extrahepatic lesions that are too small to characterize or biopsy are eligible.
* Second primary malignancy, except for adequately treated non-melanoma skin cancer, or other malignancy treated at least 3 years previously without evidence of recurrence or with a life expectancy longer than 5 years.
* Known homozygous dihydropyrimidine dehydrogenase (DPYD) deficiency
* Prior hepatic radiation, ablation, or resection for iCCA.
* Clinical evidence of portal hypertension (ascites, gastroesophageal varices, or portal vein thrombosis). Some postoperative ascites is allowed.
* (Partial) portal vein thrombosis in future liver remnant.
* Pregnant or lactating women.
* History of psychiatric disability judged by the investigator to be clinically significant, precluding informed consent or interfering with compliance for HAIP chemotherapy.
* Serious concomitant systemic disorders that would compromise the safety of the patient or his/her ability to complete the study, at the discretion of the investigator.
* Organ allografts requiring immunosuppressive therapy.
* Serious infections (uncontrolled or requiring treatment).
* Participation in another interventional study for iCCA with survival as outcome.
* Participation in another prospective study with an interventional medical product.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Two-year hepatic recurrence free survival (hRFS) | From pump implantation until 2 years after that surgery
  The percentage of patients who do not have return of disease in the liver two years after surgery. The time frame is defined as the period between pump implantation and return of disease in the liver. A recurrence is defined as a biopsy-proven recurrent lesion or radiological evidence with cross-sectional imaging in combination with an elevated CA19.9 or CEA level in the blood samples.

SECONDARY OUTCOMES:
Overall recurrence free survival (RFS) | From pump implantation until the earliest return of disease in the body during the study (up to 5 years after inclusion)
  The percentage of patients who do not have return of disease in the given time frame. A recurrence is defined as a biopsy-proven recurrent lesion or radiological evidence with cross-sectional imaging in combination with an elevated CA19.9 or CEA level in the blood samples.
Overall survival (OS) | From pump implantation until death or lost to follow-up during the study (up to 5 years after inclusion)
  OS is defined as the interval between pump implantation and the date of death (by any cause) or date of last follow-up
Post-operative complications | From pump implantation until 90 days after surgery
  All complications rated Clavien-Dindo grade 3 or higher are recorded for the first 90 days after surgery.
Chemotherapy related adverse events (AEs) | From inclusion until 4 weeks after the end of treatment with chemotherapy
  Chemotherapy related adverse events (AEs) will be collected if they are grade III or higher according to CTCAE version 5.0
Proportion of patients started with HAIP chemotherapy | From pump implantation until the first cycle of HAIP chemotherapy, on average between 4 and 16 weeks after implantation of the HAIP chemopump
  The number of patients that could receive at least 1 cycle of HAIP chemotherapy with floxuridin
Quality of life: EORTC QLQ-30 | From inclusion until 5 years after surgery
  After study inclusion and every 3 months (+/- 30 days) thereafter patients will be asked to complete the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). This validated instrument includes 30 items covering functional domains, symptom scales, and global health status. Scores range from 0 to 100, with higher scores on the global health and functional scales indicating better quality of life.
  After 1 year of follow-up, the questionnaires will be taken annually until a maximum of 5 years.
Quality of life: EQ-5D | From inclusion until 5 years after surgery
  After study inclusion and every 3 months (+/- 30 days) thereafter patients will be asked to complete the EuroQol 5-Dimension (EQ-5D) questionnaire, a standardized measure of health-related quality of life. The EQ-5D includes five dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The resulting health state is converted into an index score ranging from 0 (equivalent to death) to 1 (perfect health), though negative scores are possible.
  After 1 year of follow-up, the questionnaires will be taken annually until a maximum of 5 years.
Cost-effectiveness | From implantation of the chemo pump until 2 years after (=timeframe of the primary outcome)
  An assessment of the cost-effectiveness of HAIP chemotherapy for patients with iCCA will be made
Predictive biomarkers in the blood for efficacy of HAIP chemotherapy | From implantation of the chemo pump until 1 year after surgery or return of disease (whichever comes first)
  A total of five additional blood samples will be collected. These samples will be collected:
  * On the day of surgery before the incision is made.
  * During surgery (directly from the hepatic vein).
  * Before the start of HAIP chemotherapy.
  * After the last cycle of HAIP chemotherapy.
  * At one year after surgery or at recurrence
Predictive biomarkers from liver tissue for efficacy of HAIP chemotherapy | From resection until 25 years after (conform applicable laws)
  Additionally, tumor tissue will be collected from the removed part of the liver during the surgery. These tissue samples will be stored for further research into biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Bas Groot Koerkamp, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The decision on sharing IPD has not been made within the trial team. Once this decision is made, we will update this part.